CLINICAL TRIAL: NCT07364201
Title: A Comparison of the Effectiveness of Nicardipine and Labetalol in Controlling Hemodynamics in Postoperative Hemorrhagic Stroke Craniotomy Patients in the Intensive Care Unit
Brief Title: A Comparison of Nicardipine and Labetalol for Blood Pressure Control in Intensive Care Patients After Hemorrhagic Stroke Brain Surgery
Acronym: NIC-LAB ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Septani Anugrah Cinditya, Principal Investigator, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SACUSU2025; 1276/KEPK/USU/2025 (Other: Ethics Committee Approval For Conducting Health Research Universitas Sumatera Utara)
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hemorrhagic Strokes; Postoperative Hypertension; Hemodynamic Instability
Keywords: Hemorrhagic Stroke; Craniotomy; Nicardipine; Labetalol; Hemodynamic Control; Intensive Care Unit; Postoperative Hypertension; Blood Pressure Management
MeSH Terms: conditions — Hemorrhagic Stroke | interventions — Nicardipine; Labetalol

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in parallel to one of two intervention groups to receive either intravenous nicardipine or intravenous labetalol during postoperative intensive care unit management. Each participant receives only one study intervention, and outcomes are compared between groups.
Masking Description: No additional parties are masked beyond the participant, care provider, investigator, and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicardipine (Experimental): Participants assigned to this arm receive intravenous nicardipine for postoperative blood pressure control during intensive care unit management following craniotomy for hemorrhagic stroke.
  Interventions: Drug: Nicardipine
- Labetalol (Experimental): Participants assigned to this arm receive intravenous labetalol for postoperative blood pressure control during intensive care unit management following craniotomy for hemorrhagic stroke.
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Nicardipine — Intravenous nicardipine is administered as a continuous infusion for postoperative blood pressure control in patients admitted to the intensive care unit after craniotomy for hemorrhagic stroke. The infusion is titrated according to a standardized protocol to achieve and maintain the target systolic blood pressure range during the first 24 hours of postoperative care.
  Arms: Nicardipine
Drug: Labetalol — Intravenous labetalol is administered as a continuous infusion for postoperative blood pressure control in patients admitted to the intensive care unit after craniotomy for hemorrhagic stroke. The infusion is titrated according to a standardized protocol to achieve and maintain the target systolic blood pressure range during the first 24 hours of postoperative care.
  Arms: Labetalol

SUMMARY:
Patients with hemorrhagic stroke who undergo brain surgery (craniotomy) often experience high blood pressure after surgery. Poor blood pressure control can increase the risk of bleeding, brain injury, and other serious complications. In the intensive care unit (ICU), intravenous blood pressure medications are commonly used to keep blood pressure within a safe range.

This study aims to compare two commonly used intravenous blood pressure medications, nicardipine and labetalol, in patients who have undergone craniotomy for hemorrhagic stroke. The study will evaluate how well each medication controls blood pressure and heart rate during the first 24 hours of ICU care, as well as the speed at which the target blood pressure is achieved and the occurrence of side effects.

Participants will receive either nicardipine or labetalol according to the study protocol. Blood pressure and heart rate will be continuously monitored in the ICU as part of standard care. The results of this study are expected to help health care providers choose the most appropriate medication to achieve stable blood pressure control and improve postoperative care for patients with hemorrhagic stroke.

DETAILED DESCRIPTION:
Hemorrhagic stroke patients undergoing craniotomy are at increased risk of postoperative blood pressure elevation and hemodynamic instability, which may contribute to secondary brain injury, intracranial bleeding, and other postoperative complications. Appropriate blood pressure management in the intensive care unit (ICU) is therefore a critical component of postoperative care in this population.

Nicardipine and labetalol are intravenous antihypertensive agents commonly used for blood pressure control in neurocritical care settings. Both medications are recommended in current clinical practice; however, their hemodynamic profiles, including onset of action, stability of blood pressure control, and adverse effect patterns, differ. Evidence directly comparing these agents in the postoperative period following craniotomy for hemorrhagic stroke remains limited.

This study is a double-blind randomized clinical trial conducted in adult patients admitted to the ICU after craniotomy for hemorrhagic stroke. Eligible participants are randomly assigned to receive either intravenous nicardipine or intravenous labetalol according to a standardized treatment protocol. Hemodynamic monitoring, including systolic blood pressure, diastolic blood pressure, mean arterial pressure, and heart rate, is performed continuously using an arterial catheter as part of routine ICU management.

The primary objective of the study is to compare the effectiveness of nicardipine and labetalol in achieving and maintaining target systolic blood pressure during the first 24 hours of postoperative ICU care. Secondary objectives include comparison of time to reach target blood pressure, blood pressure variability, and the incidence of predefined adverse events such as bradycardia, hypotension, and tachycardia.

The findings of this study are expected to provide clinically relevant information regarding the comparative performance of nicardipine and labetalol for postoperative hemodynamic control in patients with hemorrhagic stroke, and to inform evidence-based blood pressure management strategies in neurocritical care practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old).
* Diagnosed with hemorrhagic stroke.
* Undergoing craniotomy for hemorrhagic stroke.
* Admitted to the intensive care unit after surgery.
* Require intravenous antihypertensive therapy for postoperative blood pressure control.
* Invasive arterial blood pressure monitoring in place.
* Written informed consent obtained from the patient or legally authorized representative.

Exclusion Criteria:

* Known hypersensitivity or contraindication to nicardipine or labetalol.
* Severe bradycardia, advanced atrioventricular block, or uncontrolled heart failure.
* History of bronchial asthma or severe chronic obstructive pulmonary disease.
* Hemodynamic instability requiring vasopressor support at enrollment.
* Pregnancy or breastfeeding.
* Participation in another interventional clinical study during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-01-03 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Hemodynamic Control | First 24 hours postoperatively in the intensive care unit
  Comparison of systolic blood pressure (SBP) control between the nicardipine and labetalol groups during the first 24 hours after craniotomy for hemorrhagic stroke, assessed using continuous invasive arterial blood pressure monitoring.

SECONDARY OUTCOMES:
Time to Achieve Target Systolic Blood Pressure | Within the first 24 hours postoperatively
  Time required to reach the target systolic blood pressure range (140-150 mmHg) after initiation of the study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Adam Malik Hospital, Haji Hospital Medan, Medan, North Sumatera, Indonesia